CLINICAL TRIAL: NCT00642109
Title: A Prospective Randomized Clinical Trial: Comparison of the Retropubic (TVT) With the Transobturator (outside-in T.O.T. Monarc or Inside-out TVT-O) Sling Operation in the Treatment of Female Stress Urinary Incontinence or Stress Dominated Mixed Urinary Incontinence
Brief Title: A Comparison of the Retropubic (TVT) With the Transobturator Sling Operation in the Treatment of Female Stress Urinary Incontinence or Stress Dominated Mixed Urinary Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: higher incidence of pain related sexual dysfunction in the TO arm
Sponsor: David Scheiner (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, David Scheiner, PI, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: slingrnd06
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TVT (Other): Tension-free Vaginal Tape (TVT)
  Interventions: Procedure: midurethral sling procedure
- TOT (Other): Transobturator Tape outside-in (TOT Monarc)
  Interventions: Procedure: midurethral sling procedure
- TVT-O (Other): Transobturator Tape inside-out (TVT-O)
  Interventions: Procedure: midurethral sling procedure

INTERVENTIONS:
Procedure: midurethral sling procedure — quality of life, voiding dysfunction

SUMMARY:
The midurethral tension-free vaginal tape (a macroporous polypropylene mesh) procedure is a well established technique for treating female stress urinary incontinence in patients with (hyper)mobile urethra. Postoperative continence rates are achieved in up to 95%. Currently, several anatomical approaches are developed and investigated to simplify this minimal invasive technique and make it safer. While the retropubic approach consists of the passage of the needles from under the midurethra up behind the pubic bone through the cavum retzii, the transobturator technique traverses the foramina obturatoria. Intraoperative complications like bladder perforation (in 4%) can be treated conservatively, while postoperative complications like voiding dysfunction (urinary outlet obstruction in up to 16% or urinary retention) are troublesome, impair the quality of life and require occasionally surgical sling release (transection of the sling). The aim of this study is to compare quality of life, postoperative voiding dysfunction, success rates and tape position after retropubic and transobturator sling procedure.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* Urodynamic stress urinary incontinence or stress dominated mixed urinary incontinence with mobile urethra
* With or without concomitant surgery for pelvic organ prolapse
* With or without hysterectomy

Exclusion criteria:

* No informed consent
* No preoperative urodynamic investigation
* Mixed urinary incontinence with predominant overactive bladder
* Recurrent stress urinary incontinence after sling procedure
* Begin of treatment of overactive bladder less then a month ago or non stable condition
* Pregnancy
* Desires future childbearing
* Concomitant incontinence procedure like intravesikal injection of Botulinumtoxin
* Preoperative postvoid residual urinary volume exceeding 100cc
* Coagulopathies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-01; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Urodynamic stress urinary incontinence measurement | December 2009

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, clinic for gynaecology, Zurich, Switzerland